CLINICAL TRIAL: NCT01636167
Title: Construction of Computerized Intraoperative Keratometer and Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, Clinical Professor, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Astigmatism
Record Dates: First submitted 2012-06-29; First posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Corneal Astigmatism; Orientation
MeSH Terms: conditions — Astigmatism; Orientation, Spatial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: computerized intraoperative keratomer — computerized intraoperative keratomer can analyze the axis of corneal astigmatism accurately as well as rapidly by self-designed software during surgery
  Other Names: Experimental: computerized intraoperative keratomer

SUMMARY:
To construct a computerized intraoperative keratometer to analyze the axis of corneal astigmatism accurately as well as rapidly by self-designed software during surgery.

DETAILED DESCRIPTION:
The study is designed to construct a computerized intraoperative keratometer to analyze the axis of corneal astigmatism accurately as well as rapidly by self-designed software during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cornea astigmatism from -1.0 D to -4.0D;

Exclusion Criteria:

* any significant corneal disease
* Other eye diseases induces impaired vision ,such as retinal detachment,keratoconus,pterygium,glaucoma,choroidal detachment,vitreous hemorrhage,congenital cataract,lens dislocation,anterior uveitis ,pupil deformation and so on;
* Previous corneal or intraocular surgery;
* Refuse surgery;

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
axis of astigmatism | day 1

SECONDARY OUTCOMES:
axis of implantation | day 1

CONTACTS AND LOCATIONS:
Overall Officials: YU A YONG, Principal Investigator — Wenzhou Medical University
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China